CLINICAL TRIAL: NCT03187262
Title: A Phase 2 Study of Daratumumab in Patients With Relapsed or Refractory Waldenström Macroglobulinemia
Brief Title: A Study of Daratumumab in Patients With Relapsed or Refractory Waldenström Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Jorge J. Castillo, MD, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-164
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Waldenström Macroglobulinemia
Keywords: Waldenström Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): * Daratumumab will be administered in three phases: Induction, consolidation and maintenance
  * During induction, participants will receive daratumumab on days 1, 8, 15 and 22 of each 28-day
  * During consolidation, daratumumab will be administered on days 1 and 15 of each 28-day cycle
  * During maintenance, daratumumab will be administered on day 1 of each 28-day cycle
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Daratumumab is a monoclonal human antibody. Daratumumab has shown the ability to slow or stop the growth of cells that have CD38 on the cell surface when tested in laboratories
  Other Names: Darzalex

SUMMARY:
This research study is studying Daratumumab as a possible treatment for Waldenström Macroglobulinemia.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved Daratumumab for this specific disease but it has been approved for other uses.

Daratumumab is a monoclonal human antibody. An antibody recognizes a specific protein and binds to it. Daratumumab binds to a protein called CD38 located on the surface of B cells like WM. Daratumumab has shown the ability to slow or stop the growth of cells that have CD38 on the cell surface when tested in laboratories.

In this research study, the investigators are evaluating the efficacy of Daratumumab as a single agent in participants with WM that has come back or has shown no response to previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenström Macroglobulinemia (Owen et al. 2003), and meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenström macroglobulinemia (Kyle et al. 2003)
* At least one previous treatment for WM with either documented disease progression or no response (stable disease) to the most recent treatment regimen
* Measurable disease, defined as presence of serum immunoglobulin M (IgM) with a minimum IgM level of >2 times the upper limit of normal of each institution is required
* Participants with symptomatic hyperviscosity or serum IgM >5,000 mg/dL to undergo plasmapheresis prior to treatment initiation
* Age ≥18 years
* ECOG performance status ≤2 (see Appendix A)
* Participants must have preserved organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 50,000/mcL
  * Hemoglobin ≥ 8 g/dL
  * Total bilirubin ≤ 1.5 mg/dL or < 2 mg/dL if attributable to hepatic infiltration by neoplastic disease
  * AST/ALT ≤ 2.5 × institutional upper limit of normal
  * EGFR ≥ 30 ml/min
* Not on any active therapy for other malignancies with the exception of topical therapies for basal cell or squamous cell cancers of the skin.
* Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or have or will have complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) while participating in the study; and 2) for at least 90 days after discontinuation from the study. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. FCBP must be referred to a qualified provider of contraceptive methods if needed. FCBP must have a negative serum pregnancy test at screening.
* Able to adhere to the study visit schedule and other protocol requirements.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, uncontrolled intercurrent illness, or psychiatric illness/social condition that would prevent study participation.
* Concurrent use of any other anti-cancer agents or treatments or any other investigational agents.
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known CNS lymphoma.
* New York Heart Association classification III or IV heart failure.
* Known history of Human Immunodeficiency Virus (HIV), active infection with Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV).
* Lactating or pregnant women.
* Grade >2 toxicity (other than alopecia) continuing from prior anti-cancer therapy.
* History of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge J Castillo, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Daratumumab: * Daratumumab will be administered in three phases: Induction, consolidation and maintenance
  * During induction, participants will receive daratumumab on days 1, 8, 15 and 22 of each 28-day
  * During consolidation, daratumumab will be administered on days 1 and 15 of each 28-day cycle
  * During maintenance, daratumumab will be administered on day 1 of each 28-day cycle
  Daratumumab: Daratumumab is a monoclonal human antibody. Daratumumab has shown the ability to slow or stop the growth of cells that have CD38 on the cell surface when tested in laboratories
Period: Induction
Arm/Group | Daratumumab
Started | 13
Completed | 7
Not Completed | 6
Not completed — Lack of Efficacy | 2
Not completed — Progressive Disease | 4
Period: Consolidation
Arm/Group | Daratumumab
Started | 7
Completed | 2
Not Completed | 5
Not completed — Progressive Disease | 5
Period: Maintenance
Arm/Group | Daratumumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daratumumab
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 69 [53 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Time Frame: 2 years
Population: Only participants who have measurable disease present at baseline, received at least one cycle of therapy, and had their disease re-evaluated were considered evaluable for response. 2 participants did not complete the first cycle of therapy and were unevaluable for the primary objective.
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Progression Free Survival
Description: Amount of time following daratumumab administration until >25% increase in serum IgM
Time Frame: 4 years
Population: Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response.
Measure: Median (Full Range); unit: months
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
months | 2 [1 to 28]

3. Secondary Outcome: Number of Participants With Complete Response
Description: A complete response is defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
Participants | 0

4. Secondary Outcome: Number of Participants With Partial Response
Description: Partial response (PR) is defined as achieving a ≥50% reduction in serum IgM levels.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
Participants | 2

5. Secondary Outcome: Number of Participants With Very Good Partial Response
Description: Very Good Partial Response (VGPR): is defined as ≥90% reduction in serum IgM levels, or normalization of serum IgM levels.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
Participants | 0

6. Secondary Outcome: Number of Participants With Minor Response
Description: Minor Response (MR): A minor response (MR) is defined 25-49% reduction in serum IgM levels.
Time Frame: 2 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab
Number analyzed (Participants) | 11
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline, throughout treatment with daratumumab, and for 30 days after last dose of daratumumab, up to 4 years
Arm/Group | Daratumumab
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=13)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Investigations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Neutropenia (Investigations) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
Leg weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Infusion reaction (General disorders) | 1 (1)
Strep salvarius bacteremia (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daratumumab (N=13)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Decreased Hearting (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Peripheral edema (General disorders) | 2 (2)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 4 (4)
Infusion related reaction (General disorders) | 5 (5)
Thrush (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline pohosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
AC joint separation (Musculoskeletal and connective tissue disorders) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramping (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Painful urination (Renal and urinary disorders) | 1 (1)
Ganglion cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Memory loss (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
PSA elevation (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Tender feeling on skin (Skin and subcutaneous tissue disorders) | 1 (1)
Toe blister (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT03187262/Prot_SAP_000.pdf